CLINICAL TRIAL: NCT02826486
Title: A Phase IIa, Multicenter, Open-label Study to Assess the Safety and Efficacy of the Combination of BL-8040 and Pembrolizumab in Patients With Metastatic Pancreatic Cancer, the COMBAT Study (KEYNOTE-202)
Brief Title: Study Assessing Safety and Efficacy of Combination of BL-8040 and Pembrolizumab in Metastatic Pancreatic Cancer Patients
Acronym: COMBAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-8040.PAC.201
Record Dates: First submitted 2016-06-21; First posted 2016-07-11 (Estimated); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — 4-fluorobenzoyl-TN-14003; pembrolizumab; Drug Therapy; irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: BL-8040 + Pembrolizumab (Keytruda®) (Experimental): BL-8040 monotherapy 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination therapy period begins following monotherapy treatment and consists of:
  * Pembrolizumab 200 mg once every three weeks.
  * Beginning on Day 10, BL-8040 three times a week
  Interventions: Drug: BL-8040; Drug: Pembrolizumab
- BL-8040 + Pembrolizumab + Chemotherapy (Experimental): BL-8040 monotherapy 1.25 mg/kg subcutaneous (SC) injections daily on days 1-5 of week 1 of treatment.
  Combination therapy period begins following monotherapy treatment and consists of:
  * IV Onivyde® 70 mg/m2 over 90 minutes followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab 200mg once every three weeks.
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing.
  Interventions: Drug: BL-8040; Drug: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: BL-8040 — BL-8040 subcutaneous (SC) injections
Drug: Pembrolizumab — Pembrolizumab will be given as a 30-minute IV infusion
  Other Names: Keytruda
Drug: Chemotherapy — • IV Onivyde® followed by IV leucovorin (LV), followed by IV fluorouracil (5-FU), every 2 weeks.
  Other Names: Onivyde / Leucovorin (LV) / Fluorouracil (5-FU)
  Arms: BL-8040 + Pembrolizumab + Chemotherapy

SUMMARY:
This study will assess the efficacy and safety of BL-8040 in combination with pembrolizumab (Keytruda®) and BL-8040/ Pembrolizumab in combination with liposomal irinotecan (Onivyde®)/5-fluorouracil/leucovorin (5-FU/LV) in subjects with metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
This will be an open-label, two-cohort, phase IIa study in subjects with metastatic pancreatic adenocarcinoma.

The study will be comprised of 2 cohorts,. Each includes approximately 40 subjects with unresectable metastatic pancreatic adenocarcinoma. Cohorts will be conducted sequentially (one after the other).

Each cohort study consists of two periods:

* Monotherapy period: One week, with BL-8040 administered daily on days 1-5.
* Combination therapy:

Cohort 1: Three-week cycles of a combination of BL-8040 administered three times a week (TIW) and pembrolizumab administered once every three weeks.

Cohort 2: Onivyde®/5-FU/LV every 2 weeks, pembrolizumab once every 3 weeks and BL-8040 twice a week.

Cohort 1: Subjects with metastatic pancreatic adenocarcinoma will be enrolled and receive BL-8040 monotherapy for five days followed by a combination treatment of BL-8040 and pembrolizumab. During the monotherapy period, eligible subjects will receive daily subcutaneous (SC) injections of BL-8040 (1.25 mg/kg) on Days 1 - 5.

From Day 8, subjects will begin a combination period consisting of treatment with SC BL-8040 TIW and pembrolizumab once every three weeks. The combination therapy will continue for up to 35 cycles of pembrolizumab approximately two years), or until progression, clinical deterioration or Early Termination, whichever comes first.

Cohort 2: Subjects with metastatic pancreatic adenocarcinoma that have progressed following first-line treatment with gemcitabine-based chemotherapy will be enrolled and receive BL-8040 monotherapy for five days followed by a combination treatment of BL-8040, pembrolizumab and chemotherapy. During the monotherapy period, eligible subjects will receive daily SC injections of BL-8040 on Days 1 - 5.

From Day 8, subjects will begin a combination period consisting of:

* IV Onivyde® followed by IV leucovorin (LV), followed by IV fluorouracil (5-FU), every 2 weeks.
* Pembrolizumab every three weeks.
* BL-8040 twice a week

The combination therapy will continue for up to 35 treatments (approximately two years), or until progression, clinical deterioration or Early Termination, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older.
2. Patients must sign a written informed consent prior to entering the study.
3. Histologically confirmed (either previously or newly biopsied) metastatic unresectable pancreatic adenocarcinoma, including with intraductal papillary mucinous neoplasm.
4. Have measurable disease (≥ 1 measurable lesion) based on Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 as determined by the site study team. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Previous treatment lines

   1. Cohort 1: Have documented objective radiographic progression after stopping treatment with first-line or further therapy, i.e. chemotherapy and or radiotherapy. Surgery not followed with neoadjuvant therapy will not be considered as first-line therapy.
   2. Cohort 2: Have documented objective radiographic progression after stopping treatment with first-line, gemcitabine-based chemotherapy. Only primary metastatic patients will be allowed to participate. Patients with previous surgery for their pancreatic cancer will not be allowed to participate.
6. Willing to submit an evaluable tumor tissue sample, preferably from a liver metastasis, unless tumor is considered inaccessible or biopsy is otherwise considered not in the subject's best interest
7. Complete resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia). If the subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
8. Eastern Cooperative Oncology Group (ECOG) status ≤1.
9. Life expectancy of at least 3 months.
10. Adequate organ function at Baseline as defined below. All laboratory assessments should be performed within 10 days of treatment initiation

    1. Hematological:

       * White blood cell (WBC) ≥ 2,500/mm^3
       * Absolute neutrophil count

         * Cohort 1: ≥ 1000 /mm^3
         * Cohort 2: ≥ 1500 /mm^3
       * Platelet count ≥ 100,000/mm^3
       * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
       * Hematocrit ≥30%
    2. Renal function:

       • Creatinine ≤1.5 x Upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate (GFR)) can also be used in place of creatinine or (CrCl) > 60 mL/min for subject with creatinine levels >1.5 x institutional ULN
    3. Hepatic function:

       * Total Bilirubin: within institutional normal ranges
       * Aspartate Aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT) and Alanine Transaminase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT): ≤2.5 x ULN OR ≤5 x ULN for subjects with liver metastases
    4. Coagulation:

       * International Normalized Ratio (INR) or PT: ≤1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
       * Activated Partial Thromboplastin Time (aPTT): ≤1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
11. Subjects must use effective contraception:

    1. Female subjects must be of non-childbearing potential or, if of childbearing potential, must have a negative urine or serum pregnancy test within 72 hours prior to taking study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible. Non-childbearing potential is defined as (by other than medical reasons):

       * ≥45 years of age and has not had menses for over 2 years
       * Amenorrhoeic for > 2 years without a hysterectomy and oophorectomy and a Follicle Stimulating Hormone (FSH) value in the postmenopausal range upon pretrial (Screening) evaluation
       * Post hysterectomy, bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation at least 6 weeks prior to Screening. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the subject must be willing to use two adequate barrier methods throughout the study, starting with the Screening visit through 120 days after the last dose of study therapy. Information must be captured appropriately within the site's source documents
    2. Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has a pancreatic tumor other than adenocarcinoma, including: acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma, Vater and periampullary duodenal or common bile duct malignancies.
2. For Cohort 2 only: subjects with a bowel obstruction.
3. Has an active infection requiring systemic therapy or has an uncontrolled infection.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions are adequately treated basal cell or squamous cell carcinoma that has undergone potentially curative therapy or carcinoma in situ of the cervix.
5. Has an underlying medical condition that would preclude study participation.
6. Has a disease that is suitable for therapy administered with curative intent.
7. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from Adverse Event (AE) due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at Baseline) from AE due to a previously administered agent .
11. An active autoimmune disease that has required systemic treatment in the 2 years preceding the study (i.e., with the use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has received transfusions of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including Granulocyte Colony Stimulating Factor (G-CSF), Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) or recombinant erythropoietin) within 4 weeks prior to study Day 1.
13. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
14. Has a history of interstitial lung disease.
15. O2 saturation < 92% (on room air).
16. For both Cohorts: Has unstable angina, new onset angina within the last 3 months, myocardial infarction within the last 6 months, and current congestive heart failure New York Heart Association Class III or higher. For Cohort 2: has ventricular arrhythmias or uncontrolled blood pressure, or severe arterial thromboembolic events less than 6 months prior to study initiation.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit through 120 days after the last dose of trial treatment. Women with a positive pregnancy test within 72 hours from Baseline.
20. Has received prior therapy with an anti-Programmed Cell Death Protein 1 (PD-1), anti-Programmed Cell Death-Ligand 1 (PD-L1), or anti-(Programmed Cell Death-Ligand 2 (PD-L2) agent or if the subject has previously participated in Merck MK-3475 clinical trials.
21. Has a positive HIV test at Screening or at any time prior to Screening. Patients without a prior positive HIV test result will undergo an HIV test at Screening, unless not permitted per local regulations.
22. Has known active Hepatitis B (defined as having a positive Hepatitis B surface antigen (HBsAg) test at Screening) or Hepatitis C (defined as having a positive Hepatitis C Virus (HCV) antibody test or a positive HCV RNA test at Screening)
23. Has known history of Chronic Hepatitis B or C
24. Has received a live vaccine within 30 days of the planned start of study therapy. Seasonal flu vaccines that do not contain live virus are permitted.
25. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or computerized tomography (CT) scan, for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to Baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
26. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
27. Cohort 2: Has clinical ascites requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abi Vainstein, MD, Study Chair — BioLineRx, Ltd.
Locations (31):
- United States (14):
  - Mayo Clinic, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMAC), Boston, Massachusetts
  - DF/HCC, Boston, Massachusetts
  - Karmanos Cancer Center, Wayne State University, Detroit, Michigan
  - Washington University of St Louis, St Louis, Missouri
  - Atlantic Medical Group, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Samsung Medical Center, Seoul, South Korea
- Spain (11):
  - Hospital General Universitario de Elche, Alicante
  - Vall d'Hebron, Barcelona
  - Gregorio Marañón Hospital, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - La Paz, Madrid
  - Hospitalario Universitario de Ourense, Ourense
  - Clinic Universidad de Navarra, Pamplona
  - University Hospital of Salamanca, Salamanca
  - Marques de Valdecilla de Santander, Santander
  - Hospital Universitari i Politècnic La Fe,, Valencia

REFERENCES:
- [Derived] Bockorny B, Semenisty V, Macarulla T, Borazanci E, Wolpin BM, Stemmer SM, Golan T, Geva R, Borad MJ, Pedersen KS, Park JO, Ramirez RA, Abad DG, Feliu J, Munoz A, Ponz-Sarvise M, Peled A, Lustig TM, Bohana-Kashtan O, Shaw SM, Sorani E, Chaney M, Kadosh S, Vainstein Haras A, Von Hoff DD, Hidalgo M. BL-8040, a CXCR4 antagonist, in combination with pembrolizumab and chemotherapy for pancreatic cancer: the COMBAT trial. Nat Med. 2020 Jun;26(6):878-885. doi: 10.1038/s41591-020-0880-x. Epub 2020 May 25. PMID 32451495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 - Total of 37 subjects were enrolled into the study at sites in Israel, South Korea and the US.
  Cohort 2 - Total of 43 subjects were enrolled into the study at sites in Israel, Spain and the US.
Groups:
- Cohort 1: BL-8040 + Pembrolizumab: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion)
  * Beginning on Day 10, BL-8040 three times a week (given as SC injections)
- Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Chemotherapy: IV Onivyde® 70 mg/m2 over 90 minutes, followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion).
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing (given by SC injections).
Period: Overall Study
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
Started | 37 | 43
Completed | 0 | 0
Not Completed | 37 | 43

BASELINE CHARACTERISTICS:
Population: Cohort 1 & Cohort 2: Full analysis set - all enrolled subjects.
Groups:
- BL-8040 + Pembrolizumab + Chemotherapy: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Chemotherapy: IV Onivyde® 70 mg/m2 over 90 minutes followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion)
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing (given by SC injections)
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | BL-8040 + Pembrolizumab + Chemotherapy | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.2) | 66.3 (9.6) | 65.35 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 18 | 24 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 33 | 36 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  South Korea | 2 | 0 | 2
  United States | 18 | 17 | 35
  Israel | 17 | 7 | 24
  Spain | 0 | 19 | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed by Imaging According to RECIST 1.1 Criteria
Description: Response is determined by assessment of target lesions identified in CT or MRI imaging.
  The ORR is assessed according to RECIST 1.1, defined as the sum of PRs (Partial Responses) and CRs (Complete Responses) determined according to best response RECIST 1.1 criteria.
  PR is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
  CR is defined as disappearance of all target lesions.
Time Frame: Change in response between screening, end of monotherapy (Day 5), end of cycle 2 (Day 28) and approximately every 63 days until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
Population: Best Response according to RECIST 1.1 Principal analysis for this endpoint used the mITT Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: BL-8040 + Pembrolizumab: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion)
  * Beginning on Day 10, BL-8040 three times a week (given as SC injections) Principal analysis for this endpoint used the mITT Analysis Set N=30
- Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Chemotherapy: IV Onivyde® 70 mg/m2 over 90 minutes, followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion).
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing (given as SC injections) Principal analysis for this endpoint used the mITT Analysis Set N=39
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 30 | 39
Participants | 1 | 8

2. Secondary Outcome: Overall Survival
Description: The length of time elapsed from monotherapy Day 1 to death
Time Frame: Through study completion, an average of 2 years for cohort of the study, and follow-up until date of death up to 100 weeks.
Population: Intention To Treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 1: BL-8040 + Pembrolizumab: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion).
  * Beginning on Day 10, BL-8040 three times a week (given as SC injections)
- Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy: Monotherapy: BL-8040 1.25 mg/kg subcutaneous (SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Chemotherapy: IV Onivyde® 70 mg/m2 over 90 minutes, followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion).
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing (given as SC injections)
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 37 | 43
months | 3.3 [2.8 to 7.5] | 6.6 [4.5 to 8.7]

3. Secondary Outcome: Progression-free Survival (PFS) by Imaging (RECIST 1.1)
Description: Progression-free Survival (PFS) by imaging (assessed according to RECIST 1.1).
  Progression is determined by assessment of target lesions identified in CT or MRI imaging. Progression is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Through study completion, an average of 2 years
Population: Intention to treat population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy: Monotherapy: BL-8040 1.25 mg/kg subcutaneous(SC) injections daily on Days 1-5 of Week 1 of treatment.
  Combination Therapy: Combination therapy period begins following monotherapy treatment and consists of:
  * Chemotherapy: IV Onivyde® 70 mg/m2 over 90 minutes, followed by IV leucovorin (LV) 400 mg/m2 over 30 minutes or according to local standard, followed by IV fluorouracil (5-FU) 2400 mg/m2 over 46 hours, every 2 weeks.
  * Pembrolizumab (Keytruda®) 200 mg once every three weeks (given as a 30 minute IV infusion).
  * Beginning on Day 10, BL-8040 twice a week and following the chemotherapy dosing (given as SC injections)
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 37 | 43
Months | 1.5 [1.5 to 1.8] | 3.8 [1.6 to 5.1]

4. Secondary Outcome: Disease Control (DC)
Description: Sum of Partial Response (PR), Complete Response (CR) and Stable Disease (SD). PR is defined as an at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
  CR is defined as disappearance of all target lesions. Progressive Disease (PD) is defined as an at least 20% increase in the sum of the longest diameter of target lesions.
  SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Through study completion, an average of 2 years
Population: Modified Intention To Treat (mITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 30 | 39
Participants | 10 | 25

ADVERSE EVENTS:
Time Frame: Study treatment duration, up to 2 years for each cohort. cohort 1 and cohort 2 were conducted sequentially, with cohort 2 initiated following completion of cohort 1
Arm/Group | Cohort 1: BL-8040 + Pembrolizumab | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 5/37 | 7/43
Serious Adverse Events (participants affected / at risk) | 27/37 | 27/43
Other Adverse Events (participants affected / at risk) | 37/37 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: BL-8040 + Pembrolizumab (N=37) | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy (N=43)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (4)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: BL-8040 + Pembrolizumab (N=37) | Cohort 2: BL-8040 + Pembrolizumab + Chemotherapy (N=43)
Anemia (Blood and lymphatic system disorders) | 7 (9) | 14 (42)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8) | 5 (10)
Palpitation (Cardiac disorders) | 3 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 2 (2) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 14 (21) | 14 (22)
Ascites (Gastrointestinal disorders) | 5 (12) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (17) | 8 (13)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 22 (70)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (5)
Flatulence (Gastrointestinal disorders) | 3 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 13 (21) | 29 (71)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (29) | 23 (72)
Asthenia (General disorders) | 5 (7) | 16 (24)
Chills (General disorders) | 6 (12) | 3 (4)
Fatigue (General disorders) | 21 (33) | 21 (58)
Injection site bruising (General disorders) | 5 (8) | 0 (0)
Injection site discomfort (General disorders) | 2 (4) | 2 (6)
Injection site erythema (General disorders) | 11 (36) | 5 (7)
Injection site haemorrhage (General disorders) | 2 (2) | 0 (0)
Injection site induration (General disorders) | 2 (3) | 4 (5)
Injection site nodule (General disorders) | 2 (3) | 1 (1)
Injection site pain (General disorders) | 22 (45) | 28 (63)
Injection site pruritus (General disorders) | 13 (15) | 5 (8)
Injection site rash (General disorders) | 4 (5) | 0 (0)
Injection site reaction (General disorders) | 8 (11) | 6 (8)
Injection site swelling (General disorders) | 5 (7) | 1 (1)
Injection site warmth (General disorders) | 2 (3) | 1 (1)
Oedema peripheral (General disorders) | 7 (9) | 7 (10)
Pain (General disorders) | 2 (3) | 3 (3)
Pyrexia (General disorders) | 8 (21) | 10 (16)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (10)
Blood alkaline phosphatase increased (Investigations) | 7 (12) | 5 (6)
Blood bilirubin increased (Investigations) | 7 (11) | 5 (5)
Blood creatinine increased (Investigations) | 2 (5) | 3 (7)
Blood glucose increased (Investigations) | 3 (7) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 5 (6)
Platelet count decreased (Investigations) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 5 (11) | 9 (20)
White blood cell count increased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 17 (22) | 18 (30)
Dehydration (Metabolism and nutrition disorders) | 6 (8) | 6 (11)
Hyperglicaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (13) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 6 (10)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (5)
Dizziness (Nervous system disorders) | 4 (4) | 9 (11)
Dysgeusia (Nervous system disorders) | 3 (3) | 8 (11)
Headache (Nervous system disorders) | 3 (4) | 5 (8)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 5 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (19) | 8 (11)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (68) | 15 (44)
Rash (Skin and subcutaneous tissue disorders) | 12 (19) | 12 (25)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (15) | 2 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (29) | 2 (11)
Flushing (Vascular disorders) | 14 (27) | 7 (29)
Hypertension (Vascular disorders) | 7 (30) | 2 (47)
Hypotension (Vascular disorders) | 5 (10) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (7)
Vision blurred (Eye disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 4 (4)
Mucosal inflammation (General disorders) | 0 (0) | 6 (10)
Oedema (General disorders) | 0 (0) | 3 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hypothyroidism (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (8)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (14)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restrictions are as per the signed agreement with each PI and institution.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT02826486/Prot_SAP_000.pdf